CLINICAL TRIAL: NCT04663919
Title: Comparison of the Effects of Weight Changes on Serum Adipokines in Patients Diagnosed With Anorexia Nervosa and Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Turker, MD, PhD; Academivian; Principle Investigator, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 246164
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Anorexia Nervosa; Bariatric Surgery; Weight Change, Body
Keywords: adipocytokines; leptin; adiponectin; omentin; apelin; IL-6; Anorexia Nervosa; Bariatric Surgery; fat mass
MeSH Terms: conditions — Anorexia Nervosa; Body Weight Changes | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anorexia Nervosa (Active Comparator): Patients diagnosed with Anorexia Nervosa, having a BMI of <18, being followed up and treated in the Psychiatry Eating Disorders Polyclinic and endocrinology outpatient clinics, and who have approximately 10% weight gain during the treatment process
  Interventions: Behavioral: Dietary intervention
- Morbidly Obese (Active Comparator): Patients with a BMI> 40 diagnosed with Morbid Obesity and who lost approximately 10% of their weight by performing obesity surgery (gastric bypass or sleeve gastrectomy)
  Interventions: Procedure: Bariatric surgery-RYGB
- Healthy Volunteer (No Intervention): Volunteers with normal BMI and without any additional chronic disease

INTERVENTIONS:
Procedure: Bariatric surgery-RYGB — After the creation of a 15-25-cc gastric pouch from the upper stomach, transection of proximal jejunum 70 cm from Treitz ligament also called "alimentary tract" and anastomosis of the distal end of jejunum to the gastric pouch, and thereafter, anastomosis of the proximal end of transected jejunum to the distal part of the jejunum at 150 cm below the site of transection (jejunoileal anastomosis).
  Arms: Morbidly Obese
Behavioral: Dietary intervention — High-calorie medical nutrition program to ensure weight gain
  Arms: Anorexia Nervosa

SUMMARY:
In this study, when patients diagnosed with AN started treatment and their weight increased by 10%; On the other hand, it was aimed to compare the changes in serum adipokine levels observed in morbidly obese patients before bariatric surgery and when they lost 10% of their post-op weight with both anthropometric measurements, biochemical parameters, and values of healthy volunteers.

DETAILED DESCRIPTION:
The most characteristic feature of obesity is the increase in adipose tissue. On the contrary, in anorexia nervosa, there is a decrease in adipose tissue enough to impair neuroendocrine functions. Adipose tissue is formed by loosely binding lipid-filled cells called adipocytes and is now considered an important part of energy metabolism. Adipokines it secretes play a role in many physiological processes of the body such as nutrition, appetite, energy balance, insulin, and glucose metabolism, lipid metabolism, regulation of blood pressure, vascular remodeling, coagulation, and inflammation.

Therefore, changes in the amount of body fat in these two patient groups, which are at the two ends of the spectrum, affect both the biochemical parameters and physiological functions of the patients in different ways. It is expected that both adipokine levels and biochemical parameters will approach the values of healthy subjects with a decrease in adipose tissue of clinically morbidly obese patients and an increase in adipose tissue of patients with AN. However, in some studies comparing the parameters of patients with constitutionally weak patients and patients with AN, results contrary to expectations were obtained. In this study, we compared the extent to which weight changes changed adipokines and correlated with biochemical parameters based on healthy and normal-weight volunteers.

ELIGIBILITY:
Inclusion Criteria:

* for Anorexia Nervosa group:

  * Have been diagnosed with anorexia nervosa
  * BMI <18 kg/m2
  * Good general health
  * Volunteering to participate in the study
* for Morbidly Obese group:

  * Who was diagnosed with morbid obesity and planned to undergo RYGB operation
  * BMI> 40 kg/m2
  * Volunteering to participate in the study
* for Healthy Volunteers:

  * Good general health
  * BMI >20 and <30 kg/m2
  * Volunteering to participate in the study

Exclusion Criteria:

* <13 and> 60 years old
* to had type 2 diabetes, hypertension, liver and kidney failure, cancer, or a chronic disease

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-04-07 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Plasma Leptin levels changes: | 3 months on average
  Change in baseline Leptin levels at when decreasing by 10 percent or increasing by 10 percent from initial weight. Measured by plasma samples.
Plasma Apelin levels changes | 3 months on average
  Change in baseline Apelin levels at when decreasing by 10 percent or increasing by 10 percent from initial weight. Measured by plasma samples.
Plasma Omentin levels changes | 3 months on average
  Change in baseline Omentin levels at when decreasing by 10 percent or increasing by 10 percent from initial weight. Measured by plasma samples.
Plasma Adiponectin levels changes | 3 months on average
  Change in baseline Adiponectin levels at when decreasing by 10 percent or increasing by 10 percent from initial weight. Measured by plasma samples.
Plasma IL-6 levels changes | 3 months on average
  Change in baseline IL-6 levels at when decreasing by 10 percent or increasing by 10 percent from initial weight. Measured by plasma samples.

SECONDARY OUTCOMES:
Weight change | 3 months on average
  Change in baseline weight (kg) at when decreasing by 10 percent or increasing by 10 percent from initial weight.
Fat mass change | 3 months on average
  Change in baseline fat mass (kg) at when decreasing by 10 percent or increasing by 10 percent from initial weight.
Fat free mass changes | 3 months on average
  Change in baseline fat free mass (kg) at when decreasing by 10 percent or increasing by 10 percent from initial weight.

OTHER OUTCOMES:
Serum glucose change | 3 months on average
  Change in baseline glucose (mg/dl) at when decreasing by 10 percent or increasing by 10 percent from initial weight.
Serum insulin change | 3 months on average
  Change in baseline insulin (µU/mL) at when decreasing by 10 percent or increasing by 10 percent from initial weight.
Serum CRP change | 3 months on average
  Change in baseline CRP at when decreasing by 10 percent or increasing by 10 percent from initial weight.